CLINICAL TRIAL: NCT05742425
Title: The Efficacy and Safety of Serplulimab Combined With FOLFIRI and Bevacizumab in the Treatment of pMMR/Ras/BRAF Wild-type Unresectable Colon Cancer Peritoneal Metastases: a Multicenter Single-arm Phase II Trial
Brief Title: Serplulimab Combined With FOLFIRI and Bevacizumab in the Treatment of Colon Cancer Peritoneal Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Changxing People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1000
Record Dates: First submitted 2023-02-05; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Unresectable Colon Cancer Peritoneal Metastases; PMMR/Ras/BRAF Wild-type
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One-arm research group (Experimental)
  Interventions: Drug: Serplulimab Combined With FOLFIRI and Bevacizumab

INTERVENTIONS:
Drug: Serplulimab Combined With FOLFIRI and Bevacizumab — For patients with confirmed failure to reach CC0/1, they should be treated with sullizumab combined with FOLFIRI+bevacizumab for 4-8 cycles within 3 weeks after the exploration operation. After the end of the 4th and 8th cycles, they should be evaluated with imaging and MDT. If the conversion is successful, they should be treated with a second exploration operation within 3-4 weeks, The patients with CC0/1 can be evaluated for tumor reduction surgery (CRS) combined with intraperitoneal hyperthermic perfusion chemotherapy (HIPEC), and the follow-up treatment plan will be selected according to the clinical situation of the patients after surgery; If CC0/1 cannot be evaluated after the second exploration surgery and CC0/1 cannot be performed after the imaging evaluation, other chemotherapy and optimal supportive treatment will be performed according to the situation.

SUMMARY:
Multicentric randomised trial. The goal of this clinical research study is to evaluate the efficacy and safety of serplulimab combined with FOLFIRI+bevacizumab in the treatment of pMMR/Ras/BRAF wild-type unresectable peritoneal metastasis of colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Colon cancer was confirmed by histology, and its gene detection was pMMR/MSS and RAS/BRAF wild-type. Imaging showed peritoneal metastasis.
* 2. Peritoneal metastatic carcinoma that could not reach CC0/1 was detected surgically.
* 3. Patients with the following general characteristics:

  1. Age between 18 and 75 years
  2. Performance Status (ECOG) 0, 1 or 2, life expectancy > 12 weeks
  3. Adequate renal, and bone marrow function: a. Leukocytes >/= 3,000/microL; b. Absolute neutrophil count >/= 1,500/microL; c. Platelets >/= 100,000/Ul; d. Serum creatinine </= 1.5 mg/dL
* 4. Hepatic function: AST (SGOT)/ALT (SGPT) </= 5 X institutional (Upper Limit of Normal) ULN.
* 5. Able to tolerate immunotherapy, chemotherapy and surgery.
* 6. Patients will be informed and a signed consent before initiating any procedure specific to the trial.

Exclusion Criteria:

* 1. Age >75years or age<18years.
* 2. Cancers of non colonic origin.
* 3. History of cancer (excepted cutaneous basal cell carcinoma or in situ carcinoma of the uterine cervix) with a recurrence during the 5 previous years.
* 4. Known HIV, Hepatitis B or Hepatitis C positive.
* 5. Pregnant women or likely to be pregnant.
* 6. Persons under guardianship.
* 7. Subjects deemed unable to comply with study and/or follow-up procedures.
* 8. Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  The period from the beginning of treatment to the first occurrence of disease progression or death from any cause. If such situation is not met, the last evaluation date shall be used for analysis. In addition, if the treatment is terminated without confirming the progress of the disease, the imaging examination and follow-up should also be carried out after the treatment is terminated.

SECONDARY OUTCOMES:
Objective Remission Rate (ORR) | 3 months after preoperative chemotherapy
  The proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit. The remission period usually refers to the period from the beginning of curative effect to the confirmation of tumor progression. The objective response rate is generally defined as the sum of complete response plus partial response (CR+PR).
3-year overall survival (OS) | 3 years
  The time from the date of treatment to the date of death due to any reason. For patients who survived in the final analysis, the date of the last contact will be recorded.
CC0/1 resection rate | during operation
  Complete tumor reduction surgery: CC-0: no peritoneal residual tumor; CC-1: residual tumor diameter<2.5mm.
Incidence rate of adverse events | Baseline before any treatment,3 months after any treatment
  According to NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lifeng Sun, Principal Investigator — Zhejiang University
Locations (1):
- Changxing County People's Hospital, Huzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No